CLINICAL TRIAL: NCT07180420
Title: Proof of Concept (PoC) Evaluation of Naloxone Unique Intramuscular (IM) Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: STAT Therapeutics Inc (Industry)
Collaborators: Johnson County ClinTrials (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAT501-01
Record Dates: First submitted 2025-09-05; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer - Complete
Keywords: naloxone intramuscular forearm

STUDY DESIGN:
Intervention Model Description: The study was an outpatient, open-label, single period, single treatment, single dose proof of concept (PoC) trial in 12 healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Naloxone intramuscular (IM) (Experimental): intramuscular (IM) to extensor digitorum communis (EDC)/forearm muscle
  Interventions: Drug: naloxone IM

INTERVENTIONS:
Drug: naloxone IM — naloxone IM to the EDC/forearm muscle

SUMMARY:
WHAT IS THE PURPOSE OF THIS RESEARCH STUDY

This research study is designed to demonstrate that intramuscular (IM) Injection of FDA Approved Naloxone Hydrochloride (HCI) given in the forearm muscle is approximately the same as given the injection in the buttocks muscle. STAT Therapeutics Inc. is sponsoring this research study.

BACKGOUND AND PURPOSE FOR THIS STUDY

You are being asked to participate in this research study because you are between the ages of 18 and 55 and appear to be in stable health. Naloxone HCI is FDA approved and has been used to treat symptoms of opioid overdose for over 40 years. This research study is designed to demonstrate that intramuscular (IM) Injection of FDA Approved Naloxone Hydrochloride (HCI) given in the forearm is approximately the same as given the injection in the buttocks.

This is the first time Naloxone Hydrochloride (HCI) is given in the forearm muscle.

This is an open-label study. This means that you, the Doctor, study staff, and the Sponsor will know the study drug and the dose that you are given.

DETAILED DESCRIPTION:
WHAT IS THE PURPOSE OF THIS RESEARCH STUDY

This research study is designed to demonstrate that intramuscular (IM) Injection of FDA Approved Naloxone Hydrochloride (HCI) given in the forearm muscle is approximately the same as given the injection in the buttocks muscle. STAT Therapeutics Inc. is sponsoring this research study.

BACKGOUND AND PURPOSE FOR THIS STUDY

You are being asked to participate in this research study because you are between the ages of 18 and 55 and appear to be in stable health. Naloxone HCI is FDA approved and has been used to treat symptoms of opioid overdose for over 40 years. This research study is designed to demonstrate that intramuscular (IM) Injection of FDA Approved Naloxone Hydrochloride (HCI) given in the forearm is approximately the same as given the injection in the buttocks.

This is the first time Naloxone Hydrochloride (HCI) is given in the forearm muscle.

This is an open-label study. This means that you, the Doctor, study staff, and the Sponsor will know the study drug and the dose that you are given.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years of age
* Body mass index (BMI) 18 to 30 kg/m2
* Subjects who do not take prescribed or OTC medications on a regular basis. In the case of recent sporadic use for minor illness, the subject may be enrolled if the investigator deems the use insignificant to study.
* Nonsmokers and subjects who smoked 10 or fewer cigarettes per day.
* Be willing to spend at least 12 hours in the study facility.

Exclusion Criteria:

* Subjects who do not fulfill criteria as described in Inclusion Criteria above
* Abnormal wrist or forearm anatomy (or history of prior wrist/forearm surgery).
* Difficult venous access for blood draws
* Active infection in including respiratory tract infection
* Used opioid analgesics for pain relief within the previous 14 days, or, in the judgment of the investigator, had significant acute or chronic medical conditions.
* Known previous or concomitant serious illness or medical condition such as malignancy, HIV, significant gastrointestinal or hepatic disease or cardiovascular event or hepatitis that in the opinion of the investigator may interfere with participation in the study
* Previous Substance Use Disorder (SUD) with injectable drugs.
* Compromised cardiovascular system (history of myocardial infarction- MI, angina, etc., at discretion of principal investigator- PI).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-03-24 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Profile (area under the curve AUC) | 1 day
  Area under the Curve (AUC)

SECONDARY OUTCOMES:
PK Profile (Cmax, Tmax, T/2- half-life) | 1 day
  Pharmacokinetic (PK) profile to include (area under the curve (AUC), maximum plasma concentration (Cmax), time to maximum plasma concentration (Tmax) and half life (T/2))

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Krol, PharmD, Study Chair — STAT Therapeutics Inc
Locations (1):
- JCCT, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Healthy volunteers